CLINICAL TRIAL: NCT01001832
Title: A Phase II/III, Multicenter, Randomized, Double-Blind, Double-Dummy Study to Assess Similarity of the Efficacy, Pharmacokinetics, Safety and Immunogenicity of Abatacept Administered Subcutaneously or Intravenously in Japanese Subjects With Rheumatoid Arthritis, Receiving Background Methotrexate, and Experiencing an Inadequate Response to Methotrexate
Brief Title: Efficacy, Pharmacokinetics, Safety, and Immunogenicity Study of Abatacept Administered Subcutaneously to Treat Rheumatoid Arthritis in Japanese Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-250
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous (SC) abatacept, 125 mg (Active Comparator)
  Interventions: Drug: Subcutaneous (SC) abatacept
- Intravenous (IV) abatacept, 125 mg (Active Comparator)
  Interventions: Drug: Intravenous (IV) abatacept

INTERVENTIONS:
Drug: Intravenous (IV) abatacept — IV vial, 125-mg infusions on Days 1, 15, and 29, and every 28 days thereafter until Day 141.
  Other Names: BMS-188667
  Arms: Intravenous (IV) abatacept, 125 mg
Drug: Subcutaneous (SC) abatacept — Solution in prefilled syringes, SC, 125 mg, once weekly, for 169 days and then for 52 weeks
  Other Names: BMS-188667
  Arms: Subcutaneous (SC) abatacept, 125 mg

SUMMARY:
The purpose of this study is to assess the efficacy, pharmacokinetics, safety, and immunogenicity of abatacept after subcutaneous and intravenous administration in Japanese participants with active rheumatoid arthritis and inadequate response to methotrexate.

ELIGIBILITY:
Key Inclusion Criteria:

* Meeting criteria of the American Rheumatism Association for the diagnosis of rheumatoid arthritis (RA) and the American College of Rheumatology functional Classes I, II, or III.
* Inadequate response (as deemed by investigator) to methotrexate taken for at least 3 months (12 weeks) at a stable dose (6 to 8 mg/week) for 28 days prior to randomization (Day 1).
* Stabilization requirements for concomitant therapy: Oral corticosteroid treatment reduced to the equivalent of ≤10 mg prednisolone daily for 28 days and stabilized for at least 25 of 28 days prior to treatment (Day 1). No intra-articular, intravenous, or intramuscular injections of corticosteroids were permitted within 28 days prior to randomization (Day 1.)
* Washout requirements: Participants receiving combination RA therapy had to discontinue the following therapies at least 28 days prior to treatment (Day 1):

disease-modifying antirheumatic drugs (DMARDs), such as gold (auranofin and aurothiomalate sodium), actarit, bucillamine, azathioprine, salazosulfapyridine, lobenzarit disodium, D-penicillamine, cyclophosphamide, mycophenolate mofetil, mizoribine; cyclosporin, tacrolimus, and other calcineurin inhibitors; and immunoadsorption columns.

* Disease Activity Requirements: At randomization (Day 1), participants had to meet the following disease activity criteria: Swollen joint count: 10 or more swollen joints (66 joint count); tender joint count: 12 or more tender joints (68 joint count); C reactive protein (CRP): ≥0.8 mg/dL (result from screening visit).
* For participants receiving methotrexate plus other DMARDs(washout of a combination therapy required): At screening visit, participants had to meet the following disease activity criteria: Swollen joint count: 6 or more swollen joints (66 joint count); tender joint count: 8 or more tender joints (68 joint count); CRP: no restriction on CRP (not applicable).
* After washout, at randomization (Day 1), participants must meet the following disease activity criteria: Swollen joint count-10 or more swollen joints (66 joint count) and tender joint count-12 or more tender joints (68 joint count) and CRP: ≥0.8 mg/dL (result from screening visit). For those whose screening period were longer than 4 weeks, CRP test needed to be performed on Day
* 28 to Day -3 (prior to treatment Day 1) to verify eligibility.

Key Exclusion Criteria:

* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease. Concomitant medical conditions that, in the opinion of the investigator, might place the participant at unacceptable risk for participation in this study.
* Female participants who had undergone breast cancer screening that was suspicious for malignancy, and in whom the possibility of malignancy could not be reasonably excluded following additional clinical, laboratory, or other diagnostic evaluations.
* History of cancer within the last 5 years (other than nonmelanoma skin cell cancers cured by local resection)
* Existing nonmelanoma skin cell cancers had been removed prior to the first administration. Participants with carcinoma in situ, treated with definitive surgical intervention prior to study entry were allowed to participate.
* Clinically significant drug or alcohol abuse
* Any serious acute bacterial infection (such as pneumonia or pyelonephritis unless treated and completely resolved with antibiotics)
* Serious, chronic, or recurrent bacterial infections (such as recurrent pneumonia, chronic bronchiectasis)
* Those at risk for tuberculosis (TB). Specifically, those with current clinical, radiographic, or laboratory evidence suggestive of active TB; history of active TB within the last 3 years, even if treated; history of active TB more than 3 years ago unless there was documentation that the prior anti-TB treatment was appropriate in type and duration; latent TB that was not successfully treated. Participants with a positive result on TB screening test indicative of latent TB were not eligible for the study unless active TB infection had been ruled out and treatment for latent TB with isoniazid had been initiated for at least 4 weeks prior to administration of the study drug and the participant had a negative finding for TB on a chest X-ray film at enrollment.
* Herpes zoster resolving less than 2 months prior to enrollment
* Current evidence (as assessed by the investigator) suggestive of active or latent bacterial or viral infections, including human immunodeficiency virus infection.
* Physical examination and laboratory test findings: Hepatitis B surface antigen-positive status; hepatitis C antibody-positive status. Any of the following laboratory values: Hemoglobin concentration: <.5 g/dL; white blood cell count: <3,000/μL (3*10^9/L); platelet count: <100,000/mm^3(100*10^9/L); serum creatinine: >2 times upper limit of normal (ULN); serum alanine aminotransferase: >2 ULN; serum aspartate aminotransferase: >2 ULN.
* Prohibited treatments and/or therapies: Prior exposure to abatacept (CTLA4-Ig); prior RA treatment with any biologics, such as anti-tumor necrosis factor therapy; prior exposure to any investigational biologic not currently approved in Japan; exposure to any study medication in any other previous study within 4 weeks or 5 half-lives, whichever was longer; receipt of any live vaccines within 3 months of administration of study medication or scheduled to receive live vaccines.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- Japan (29):
  - Local Institution, Narita-Shi, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu-Shi, Fukuoka
  - Local Institution, Kurume-Shi, Fukuoka
  - Local Institution, Maebashi, Gunma
  - Local Institution, Takasaki-Shi, Gunma
  - Local Institution, Higashi-Hiroshima-Shi, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanzaki-Gun, Hyōgo
  - Local Institution, Kato-Shi, Hyōgo
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Hitachi-Shi, Ibaraki
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Sagamihara-Shi, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Nagano, Nagano
  - Local Institution, Kurashiki-Shi, Okayama-ken
  - Local Institution, Hannan-Shi, Osaka
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Kawagoe-Shi, Saitama
  - Local Institution, Kitamoto-Shi, Saitama
  - Local Institution, Tokorozawa-Shi, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Shizuoka, Shizuoka
  - Local Institution, Shimotsuke-Shi, Tochigi
  - Local Institution, Utsunomiya, Tochigi
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Nakano-Ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo

REFERENCES:
- [Derived] Amano K, Matsubara T, Tanaka T, Inoue H, Iwahashi M, Kanamono T, Nakano T, Uchimura S, Izumihara T, Yamazaki A, Karyekar CS, Takeuchi T; Japan Abatacept Study Group. Long-term safety and efficacy of treatment with subcutaneous abatacept in Japanese patients with rheumatoid arthritis who are methotrexate inadequate responders. Mod Rheumatol. 2015 Sep;25(5):665-71. doi: 10.3109/14397595.2015.1012786. PMID 25698370
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started 8 December 2009; short-term period ended 25 February 2011; long-term period ended 26 October 2012.
Pre-assignment Details: 171 participants were enrolled, 118 participants were randomized and treated in the short-term period.
Groups:
- Subcutaneous (SC) Abatacept, 125 mg: Short-term period: Participants received SC abatacept, 125 mg, injections weekly, after an intravenous (IV) abatacept loading dose on Day 1, based on body weight. Participants also received SC injections of placebo, with a loading dose of IV abatacept (and not IV placebo) administered on Day 1.
  Long-term period: All participants received weekly SC abatacept, 125 mg, for 1 year (52 weeks) without any IV infusions (active or placebo).
  Follow-up period was up to 168 days after the last dose of drug.
- Intravenous (IV) Abatacept, 125 mg: Short-term period: Participants received IV abatacept, 125 mg, infusions on Days 1, 15, and 29, and every 28 days thereafter until Day 141. Participants also received subcutaneous (SC) injections of placebo.
  Long-term period: All participants received weekly SC abatacept, 125 mg, for 1 year (52 weeks) without any IV infusions (active or placebo).
  Follow-up period was up to 168 days after the last dose of drug.
Period: Short-term Period
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Started | 59 | 59
Completed | 57 | 56
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 3
Period: Long-term Period
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Started | 56 (1 participant completed the short term period but discontinued before start of the Long-term Period.) | 56
Completed | 52 | 51
Not Completed | 4 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Other | 1 | 2
Period: Follow-up Period
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Started | 52 | 51
Completed | 34 | 30
Not Completed | 18 | 21
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Follow-up no longer required /protocol | 15 | 20
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (12.3) | 55.2 (13.6) | 55.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 48 | 86
  Male | 21 | 11 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 58 | 59 | 117
  Asian (not Japanese) | 1 | 0 | 1
Duration of Disease [Mean (Standard Deviation); unit: Years] | 7.5 (9.2) | 5.3 (7.3) | 6.4 (8.3)
Duration of Disease Category [Number; unit: Participants]
  <= 2 years | 25 (42.4) | 30 (50.8) | 55 (46.6)
  >2 to <= 5 years | 7 (11.9) | 11 (18.6) | 18 (15.3)
  >5 to <= 10 years | 10 (16.9) | 6 (10.2) | 16 (13.6)
  >10 years | 17 (28.8) | 12 (20.3) | 29 (24.6)
Tender Joint Count [Mean (Standard Deviation); unit: Number of joints] — The number of joints the participant finds painful (tender) is counted by the investigator.
  Number of joints | 20.9 (9.3) | 22.3 (9.9) | 21.6 (9.6)
Swollen Joint Count [Mean (Standard Deviation); unit: Number of joints] — the number of the participants' joints that the investigator observes is swollen.
  Number of joints | 16.4 (7.0) | 17.6 (7.2) | 17.0 (7.1)
DAS28-CRP [Mean (Standard Deviation); unit: Units on a scale] — The Disease Activity Score 28 using C-Reactive Protein (DAS28-CRP) is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). These measures are then fed into a complex mathematical formula to produce the overall DAS (greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
  Units on a scale | 5.62 (0.84) | 5.95 (0.91) | 5.79 (0.89)
HAQ Score [Mean (Standard Deviation); unit: Units on a scale] — The Health Assessment Questionnaire(HAQ) Disability Index (DI) assesses patients' functional ability by rating their abilities over the previous week. At least 2 questions are asked from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3.
  Units on a scale | 1.28 (0.690) | 1.32 (0.64) | 1.30 (0.66)
Methotrexate dose [Mean (Standard Deviation); unit: mg/week] — The methotrexate dose is the calculated weekly total dose in the week ending at the first dose date of the Short-term Period.
  mg/week | 7.3 (1.0) | 7.3 (1.0) | 7.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Day 169 in Short Term Period
Description: The ACR score of 20 indicates the degree of improvement in a patient's rheumatoid arthritis (RA), based on ACR guidelines (ACR20). The ACR score represents a percentage. To qualify for an ACR20 score, the patient must have >=20% fewer tender joints and >=20% fewer swollen joints and show 20% improvement in at least 3 of: patient overall assessment of his/her RA, physician global assessment of the patient's RA, patient self-assessment of pain, patient self-assessment of physical functioning, and results of an erythrocyte sedimentation rate or C-reactive protein test (to assess inflammation). Percentage is calculated n/N with n=number of participants with ACR score of 20 and N= all randomized participants who received at least one dose of study drug.
Time Frame: Day 169
Population: N= All randomized participants who received at least 1 dose of study medication and were analyzed. n=number of participants with ACR20 response at Day 169: 54, 49, respectively. n/N= percentage: 54/59; 49/59.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Subcutaneous (SC) Abatacept, 125 mg: Short-term period: Participants received SC abatacept, 125 mg, injections weekly, after an intravenous (IV) abatacept loading dose on Day 1, based on body weight. Participants also received SC injections of placebo, with a loading dose of IV abatacept (and not IV placebo) administered on Day 1.
  Long-term period: All participants received weekly SC abatacept, 125 mg, for 1 year (52 weeks) without any IV infusions (active or placebo).
- Intravenous (IV) Abatacept, 125 mg: Short-term period: Participants received IV abatacept, 125 mg, infusions on Days 1, 15, and 29, and every 28 days thereafter until Day 141. Participants also received subcutaneous (SC) injections of placebo.
  Long-term period: All participants received weekly SC abatacept, 125 mg, for 1 year (52 weeks) without any IV infusions (active or placebo).
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Percentage of participants | 91.5 [81.3 to 97.2] | 83.1 [71.0 to 91.6]

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50 (ACR50) and American College of Rheumatology 70 (ACR70) Responses at Day 169 in Short Term Period
Description: The American College of Rheumatology (ACR) scores of 50 and 70 indicates the degree of improvement in a patient's rheumatoid arthritis (RA), based on ACR guidelines. The ACR score represents a percentage. To qualify for an ACR50 or ACR70 scores, the patient must have >=50% or >=70%, respectively, fewer tender joints and >=50% or >=70%, respectively, fewer swollen joints and show 50% or 70%, respectively, improvement in at least 3 of the following: patient overall assessment of his/her RA, physician global assessment of the patient's RA, patient self-assessment of pain, patient self-assessment of physical functioning, and results of an erythrocyte sedimentation rate or C-reactive protein test (to assess inflammation).
Time Frame: Day 169
Population: m= All participants who received at least 1 dose of study medication in short term period and had data available. n= participants with ACR50 or ACR70 response in the short term period. n/m= percentage
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Percentage of participants
  ACR50 (n/m=39/59, 37/59) | 66.1 [52.6 to 77.9] | 62.7 [49.1 to 75.0]
  ACR70 (n/m=22/59, 18/59) | 37.3 [25.0 to 50.9] | 30.5 [19.2 to 43.9]

3. Secondary Outcome: Mean Change From Baseline in HAQ-DI Score at Day 169 in Short Term Period
Description: Adjusted mean. The Health Assessment Questionnaire Disability Index (HAQ-DI) assesses patients' functional ability by rating their abilities over the previous week. At least 2 questions are asked from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3.
Time Frame: Baseline to Day 169
Population: All participants who received at least 1 dose of study medication were analyzed.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Units on a scale | -0.62 [-0.74 to -0.49] | -0.61 [-0.73 to -0.49]

4. Secondary Outcome: Percentage of Participants With HAQ Response at Day 169 in the Short Term Period
Description: The Health Assessment Questionnaire Disability Index (HAQ-DI) assesses patients' functional ability by rating their abilities over the previous week. At least 2 questions are asked from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3. The HAQ-DI response is defined as a reduction of at least 0.30 units in HAQ score from baseline.
Time Frame: Day 169
Population: N=All randomized participants who received at least 1 dose of study medication in short term period. n=number of participants with HAQ response in short term period; n/N=percentage of participants: 41/59 and 30/59
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Percentage of participants | 69.5 [56.1 to 80.8] | 50.8 [37.5 to 64.1]

5. Secondary Outcome: Mean Change From Baseline at Six Months in DAS28-CRP - All Treated Participants
Description: The Disease Activity Score 28 using C-Reactive Protein (DAS28-CRP) is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). An overall DAS >5.1 implies active disease; <3.2, well controlled disease; and <2.6, remission.). Baseline is Day 1 or last non-missing pre-treatment value.
Time Frame: Baseline to 6 Months
Population: All participants who received at least 1 dose of study medication with both baseline and post-baseline measurements were analyzed.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Units on a scale | -2.97 [-3.25 to -2.70] | -2.75 [-3.03 to -2.48]

6. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR)-Defined Low Disease Activity Score (LDAS) and EULAR-defined Remission (REM) at Day 169 in Short Term Period
Description: EULAR defines LDAS as DAS28-CRP less than, equal to (≤) 3.2 and defines REM as DAS28-CRP less than (<) 2.6.
Time Frame: Day 169
Population: m=All randomized participants who received at least 1 dose of study medication and with LDAS and REM data available. n= number of participants with LDAS and REM. n/m=percentage of participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 57 | 57
Percentage of participants
  LDAS (n/m= 40/57, 38/57) | 70.2 [56.6 to 81.6] | 66.7 [52.9 to 78.6]
  REM (n/m= 29/57, 23/57) | 50.9 [37.3 to 64.4] | 40.4 [27.6 to 54.2]

7. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR)-Defined Low Disease Activity Score (LDAS) and EULAR-defined Remission (REM) at Day 533 in Long Term Period
Description: EULAR defines LDAS as DAS28-CRP≤3.2 and defines REM as DAS28-CRP<2.6.
Time Frame: Day 533
Population: m=All treated participants in the long term period in the analysis with available LDAS and REM data. n=number of participants with either EULAR-defined LDAS response or EULAR-defined REM response. n/m = percentage of participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 52 | 51
percentage of participants
  LDAS (n/m= 45/52, 42/51) | 86.5 [74.2 to 94.4] | 82.4 [69.1 to 91.6]
  REM (n/m= 33/52; 32/51) | 63.5 [49.0 to 76.4] | 62.7 [48.1 to 75.9]

8. Secondary Outcome: Short-term Period: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, Discontinuations Due to SAEs, Adverse Events (AEs), Treatment-related AEs, and Discontinuations Due to AEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=related or missing relationship to study medication.
Time Frame: Baseline to Day 169
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Participants
  Deaths | 0 | 0
  SAEs | 4 | 3
  Treatment-related SAEs | 3 | 2
  Discontinuations due to SAEs | 3 | 1
  AEs | 45 | 49
  Treatment-related AEs | 31 | 35
  Discontinuations due to AEs | 3 | 3

9. Secondary Outcome: Long-term Period: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, Discontinuations Due to SAEs, Adverse Events (AEs), Treatment-related AEs, and Discontinuations Due to AEs
Description: as for outcome 8
Time Frame: Baseline to Day 533 and up to 56 days following last dose in Long-Term period
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 56 | 56
Participants
  Deaths | 1 | 0
  SAEs | 5 | 5
  Treatment-related SAEs | 4 | 3
  Discontinuation due to SAEs | 1 | 0
  AEs | 49 | 49
  Treatment-related AEs | 31 | 32
  Discontinuation due to AEs | 2 | 1

10. Secondary Outcome: Short-term Period: Number of Participants With Hematology Laboratory Values Meeting the Criteria for Marked Abnormality
Description: lower limit of normal(LLN); upper limit of normal(ULN); pretreatment(preRX). Hemoglobin (g/dL): >3 g/dL decrease from preRX; hematocrit (%): <0.75*preRX; erythrocytes (*10^6 c/uL): <0.75*preRX; platelet count (*10^9 c/uL): <0.67*LLN or >1.5*ULN, of if preRX<LLN, use 0.5*preRX and <100,000/mm^3; leukocytes (*10^3 c/uL): <0.75*LLN or >1.25*ULN, or if preRX <LLN, use <0.8*preRX or >ULN, or if preRX>ULN, use >1.2*preRX or <LLN; neutrophils+bands (*10^3 c/uL): if value <1.0*10^3 c/uL; eosinophils (*10^3 c/uL): if value >0.750*10^3 c/uL; basophils (*10^3 c/uL): if value >400/mm^3; monocytes (*10^3 c/uL): if value >2000/mm^3; lymphocytes (*10^3 c/uL): if value <0.750*10^3 c/uL or if value >7.50*10^3 c/uL.
Time Frame: Baseline to Day 169
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Participants
  Hemoglobin, low | 0 | 0
  Hemoglobin, high | NA — Not evaluated | NA — Not evaluated
  Hematocrit, low | 0 | 0
  Hematocrit, high | NA — Not evaluated | NA — Not evaluated
  Erythrocytes, low | 0 | 0
  Erythrocytes, high | NA — Not evaluated | NA — Not evaluated
  Platelet count, low | 0 | 0
  Platelet count, high | 0 | 0
  Leukocytes, low | 1 | 0
  Leukocytes, high | 2 | 3
  Neutrophils + bands (absolute), low | 1 | 0
  Neutrophils + bands (absolute), high | NA — Not evaluated | NA — Not evaluated
  Eosinophils (absolute), low | NA — Not evaluated | NA — Not evaluated
  Eosinophils (absolute), high | 1 | 2
  Basophils (absolute), low | NA — Not evaluated | NA — Not evaluated
  Basophils (absolute), high | 1 | 0
  Monocytes (absolute), low | NA — Not evaluated | NA — Not evaluated
  Monocytes (absolute), high | 0 | 0
  Lymphocytes (absolute), low | 8 | 10
  Lymphocytes (absolute), high | 0 | 0

11. Secondary Outcome: Long-term Period: Number of Participants With Hematology Laboratory Values Meeting the Marked Abnormality Criteria
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Hemoglobin (g/dL): >3 g/dL decrease from preRX; hematocrit (%): <0.75*preRX; erythrocytes (*10^6 c/uL): <0.75*preRX; platelet count (*10^9 c/uL): <0.67*LLN or >1.5*ULN, of if preRX<LLN, use 0.5*preRX and <100,000/mm^3; leukocytes (*10^3 c/uL): <0.75*LLN or >1.25*ULN, or if preRX <LLN, use <0.8*preRX or >ULN, or if preRX>ULN, use >1.2*preRX or <LLN; neutrophils+bands (*10^3 c/uL): if value <1.0*10^3 c/uL; eosinophils (*10^3 c/uL): if value >0.750*10^3 c/uL; basophils (*10^3 c/uL): if value >400/mm^3; monocytes (*10^3 c/uL): if value >2000/mm^3; lymphocytes (*10^3 c/uL): if value <0.750*10^3 c/uL or if value >7.50*10^3 c/uL.
Time Frame: Baseline to Day 533
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 56 | 56
Participants
  Hemoglobin, low | 0 | 1
  Hemoglobin, high | NA — Not evaluated. | NA — Not evaluated.
  Hematocrit, low | 0 | 0
  Hematocrit, high | NA — Not evaluated. | NA — Not evaluated.
  Erythrocytes, low | 0 | 2
  Erythrocytes, high | NA — Not evaluated. | NA — Not evaluated.
  Platelet count, low | 0 | 0
  Platelet count, high | 0 | 0
  Leukocytes, low | 0 | 2
  Leukocytes, high | 0 | 1
  Neutrophils + bands (absolute), low | 0 | 0
  Neutrophils + bands (absolute), high | NA — Not evaluated. | NA — Not evaluated.
  Eosinophils (absolute), low | NA — Not evaluated. | NA — Not evaluated.
  Eosinophils (absolute), high | 1 | 2
  Basophils (absolute), low | NA — Not evaluated. | NA — Not evaluated.
  Basophils (absolute), high | 0 | 0
  Monocytes (absolute), low | NA — Not evaluated. | NA — Not evaluated.
  Monocytes (absolute), high | 0 | 0
  Lymphocytes (absolute), low | 11 | 8
  Lymphocytes (absolute), high | 0 | 0

12. Secondary Outcome: Short-term Period: Number of Participants With Liver and Kidney Function Laboratory Values Meeting the Criteria for Marked Abnormality
Description: ULN=upper limit of normal; LLN=lower limit of normal; preRX=pretreatment. alkaline phosphatase (ALP) (U/L): >2*ULN, or if preRX>ULN, use >3*preRX; aspartate aminotransferase (AST) (U/L): >3*ULN, or if preRX>ULN, use >4*preRX; alanine aminotransferase(ALT) (U/L): >3*ULN, or if preRX>ULN, use >4*preRX; Gamma glutamyltransferase(GGT) (U/L): >2*ULN, or if preRX>ULN, use >3*preRX; bilirubin (mg/dL): >2*ULN, or if preRX>ULN, use >4*preRX; blood urea nitrogen (mg/dL): >2*preRX; creatinine (mg/dL): >1.5*preRX.
Time Frame: Baseline to Day 169
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Participants
  Alkaline phosphatase (ALP), low | NA — Not evaluated | NA — Not evaluated
  ALP, high | 0 | 0
  Aspartate aminotransferase (AST), low | NA — Not evaluated | NA — Not evaluated
  AST, high | 0 | 1
  Alanine aminotransferase (ALT), low | NA — Not evaluated | NA — Not evaluated
  ALT, high | 0 | 0
  G-glutamyl transferase (GGT), low | NA — Not evaluated | NA — Not evaluated
  GGT, high | 1 | 0
  Bilirubin, total, low | NA — Not evaluated | NA — Not evaluated
  Bilirubin, total, high | 0 | 0
  Blood urea nitrogen, low | NA — Not evaluated | NA — Not evaluated
  Blood urea nitrogen, high | 0 | 0
  Creatinine, low | NA — Not evaluated | NA — Not evaluated
  Creatinine, high | 0 | 3

13. Secondary Outcome: Short-term Period: Number of Participants With Electrolyte Laboratory Values Meeting the Criteria for Marked Abnormality
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Sodium (mEq/L): <0.95*LLN or >1.05*ULN, or if preRX<LLN, use <0.95*preRX or >ULN, or if preRX>ULN, use 1.05*preRX or <LLN; potassium (mEq/L): <0.9*LLN or >1.1*ULN, or if preRX<LLN, use <0.9*preRX or >ULN, or if preRX>ULN, use 1.1*preRX or <LLN; chloride (mEq/L): <0.75*LLN or >1.125*ULN, or if preRX<LLN, use <0.75*preRX or >ULN, or if preRX>ULN, use 1.25*preRX or <LLN; calcium (mg/dL): <0.75*LLN or >1.25*ULN, or if preRX<LLN, use <0.75*preRX or >ULN, or if preRX>ULN, use 1.25*preRX or <LLN; phosphorus (mg/dL): <0.75*LLN or >1.25*ULN, or if preRX<LLN, use <0.67*preRX or >ULN, or if preRX>ULN, use 1.33*preRX or <LLN.
Time Frame: Baseline to Day 169
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 59 | 59
Participants
  Sodium, serum, low | 0 | 0
  Sodium, serum, high | 0 | 0
  Potassium, serum, low | 0 | 0
  Potassium, serum, high | 0 | 0
  Chloride, serum, low | 0 | 0
  Chloride, serum, high | 0 | 0
  Calcium, total, low | 0 | 0
  Calcium, total, high | 0 | 0
  Phosphorus, inorganic, low | 0 | 0
  Phosphorus, inorganic, high | 0 | 0

14. Secondary Outcome: Long-term Period: Number of Participants With Liver and Kidney Function Laboratory Values Meeting the Criteria for Marked Abnormality
Description: ULN=upper limit of normal; LLN=lower limit of normal; preRX=pretreatment. ALP (U/L): >2*ULN, or if preRX>ULN, use >3*preRX; AST (U/L): >3*ULN, or if preRX>ULN, use >4*preRX; ALT (U/L): >3*ULN, or if preRX>ULN, use >4*preRX; GGT (U/L): >2*ULN, or if preRX>ULN, use >3*preRX; bilirubin (mg/dL): >2*ULN, or if preRX>ULN, use >4*preRX; blood urea nitrogen (mg/dL): >2*preRX; creatinine (mg/dL): >1.5*preRX.
Time Frame: Baseline to Day 533
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 56 | 56
Participants
  Alkaline phosphatase (ALP), low | NA — Not evaluated. | NA — Not evaluated.
  ALP, high | 0 | 0
  Aspartate aminotransferase (AST), low | NA — Not evaluated. | NA — Not evaluated.
  AST, high | 0 | 2
  Alanine aminotransferase (ALT), low | NA — Not evaluated. | NA — Not evaluated.
  ALT, high | 0 | 1
  G-glutamyl transferase (GGT), low | NA — Not evaluated. | NA — Not evaluated.
  GGT, high | 1 | 2
  Bilirubin, total, low | NA — Not evaluated. | NA — Not evaluated.
  Bilirubin, total, high | 0 | 0
  Blood urea nitrogen, low | NA — Not evaluated. | NA — Not evaluated.
  Blood urea nitrogen, high | 1 | 1
  Creatinine, low | NA — Not evaluated. | NA — Not evaluated.
  Creatinine, high | 0 | 4

15. Primary Outcome: Percentage of Participants With Sustained American College of Rheumatology (ACR) Response at Day 533 in Long Term Period - All Randomized and Treated Participants During the Long Term Period
Description: The ACR score indicates the degree of improvement in a patient's rheumatoid arthritis (RA), based on ACR guidelines. The ACR score= a percentage. To qualify for a score of 20, 50 or 70 (ACR20, ACR50 or ACR70), the patient must have >=20%, >=50% or >=70%, respectively, fewer tender joints and >=20%, >=50% or >=70%, respectively, fewer swollen joints and show 20%, 50% or 70%, respectively, improvement in at least 3 of the following: patient overall assessment of his/her RA, physician global assessment of the patient's RA, patient self-assessment of pain, patient self-assessment of physical functioning, and results of an erythrocyte sedimentation rate or C-reactive protein test (to assess inflammation). Treatment groups represent treatment received in the short term period. Percentage calculated as n/m with n=number of paticipants with sustained ACR response at Day 533; m= long term participants who received at least one dose of drug and were ACR responders in the short term period.
Time Frame: Day 533
Population: m=Long term period participants who received at least one dose of drug and were ACR responders in short term period: ACR20= 49, 46; ACR50= 35, 34; ACR70= 20, 16. n=number of paticipants with sustained ACR response at Day 533. n/m = percentage
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 49 | 46
percentage of participants
  ACR 20 (n/m= 47/49; 45/46) | 95.9 [86.0 to 99.5] | 97.8 [88.5 to 99.9]
  ACR 50 (n/m= 30/35; 32/34) | 85.7 [69.7 to 95.2] | 94.1 [80.3 to 99.3]
  ACR 70 (n/m= 15/20; 15/16) | 75.0 [50.9 to 91.3] | 93.8 [69.8 to 99.8]

16. Primary Outcome: Mean Change From Baseline in HAQ-DI Score at Day 533 in Long Term Period
Description: Adjusted mean. The Health Assessment Questionnaire Disability Index (HAQ-DI) assesses patients' functional ability by rating their abilities over the previous week. At least 2 questions are asked from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3. Treatment groups represent treatment received in the short term period. Baseline is Day 1 of the study or last non-missing pre-treatment value.
Time Frame: Baseline to Day 533
Population: Number of participants with both baseline and post-baseline measurements in HAQ-DI. Treatment groups represent treatment received in the short term period.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 52 | 51
units on a scale | -0.71 [-0.87 to -0.55] | -0.71 [-0.89 to -0.52]

17. Primary Outcome: Percentage of Participants With Health Assessment Questionnaire (HAQ) Response at Day 533 in Long Term Period
Description: The Health Assessment Questionnaire (HAQ) disability index assesses patients' functional ability by rating their abilities over the previous week. At least 2 questions are asked from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The higher the number the worse the outcome. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3. HAQ response=reduction of at least 0.30 units in HAQ score from baseline. The percentage of participants with a reduction of at least 0.30 units in their HAQ score from baseline is presented. Baseline is Day 1 of the study or last non-missing pre-treatment value. Treatment groups represent treatment received in the short term period.
Time Frame: Day 533
Population: N=number of participants treated with at least 1 dose of study drug and with HAQ data available. n=number of participants with HAQ response. n/N = 41/52 and 31/51 in SC and IV arms, respectively. Treatment groups represent treatment received in the short term period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 52 | 51
percentage of participants | 78.8 [65.3 to 88.9] | 60.8 [46.1 to 74.2]

18. Primary Outcome: Mean Change in DAS28-CRP From Baseline at Day 533 in Long Term Period
Description: The Disease Activity Score 28 using C-Reactive Protein (DAS28-CRP) is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). An overall DAS >5.1 implies active disease; <3.2, well controlled disease; and <2.6, remission.). Treatment groups represent treatment received in the short term period. Baseline is Day 1 of the study or last non-missing pre-treatment value.
Time Frame: Baseline to Day 533
Population: Participants treated with at least 1 dose of study drug and who had both baseline and post-baseline measurements were analyzed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 52 | 51
units on a scale | -3.27 [-3.58 to -2.97] | -3.49 [-3.82 to -3.17]

19. Secondary Outcome: Long-term Period: Number of Participants With Electrolyte Laboratory Values Meeting the Criteria for Marked Abnormality
Description: as for outcome 13
Time Frame: Baseline to Day 533
Population: All randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Subcutaneous (SC) Abatacept, 125 mg | Intravenous (IV) Abatacept, 125 mg
Number analyzed (Participants) | 56 | 56
Participants
  Sodium, serum, low | 1 | 0
  Sodium, serum, high | 0 | 0
  Potassium, serum, low | 0 | 2
  Potassium, serum, high | 0 | 0
  Chloride, serum, low | 0 | 0
  Chloride, serum, high | 0 | 0
  Calcium, total, low | 0 | 0
  Calcium, total, high | 0 | 0
  Phosphorus, inorganic, low | 0 | 0
  Phosphorus, inorganic, high | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to 6 months post last dose
Groups:
- Abatacept Long-term (LT) SC 125 mg: Long-term period: All participants received weekly SC abatacept, 125 mg, for 1 year (52 weeks) without any IV infusions (active or placebo). Follow-up was up to 168 days after the last dose of drug.
- Short Term Intravenous (IV) Abatacept, 125 mg: Short-term period: Participants received IV abatacept, 125 mg, infusions on Days 1, 15, and 29, and every 28 days thereafter until Day 141. Participants also received subcutaneous (SC) injections of placebo.
- Short Term Subcutaneous (SC) Abatacept, 125 mg: Short-term period: Participants received SC abatacept, 125 mg, injections weekly, after an intravenous (IV) abatacept loading dose on Day 1, based on body weight. Participants also received SC injections of placebo, with a loading dose of IV abatacept (and not IV placebo) administered on Day 1.
Arm/Group | Abatacept Long-term (LT) SC 125 mg | Short Term Intravenous (IV) Abatacept, 125 mg | Short Term Subcutaneous (SC) Abatacept, 125 mg
Serious Adverse Events (participants affected / at risk) | 10/112 | 3/59 | 4/59
Other Adverse Events (participants affected / at risk) | 68/112 | 35/59 | 25/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept Long-term (LT) SC 125 mg (N=112) | Short Term Intravenous (IV) Abatacept, 125 mg (N=59) | Short Term Subcutaneous (SC) Abatacept, 125 mg (N=59)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Medical device complication (General disorders) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept Long-term (LT) SC 125 mg (N=112) | Short Term Intravenous (IV) Abatacept, 125 mg (N=59) | Short Term Subcutaneous (SC) Abatacept, 125 mg (N=59)
Alanine aminotransferase increased (Investigations) | 9 | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 4
Periodontitis (Gastrointestinal disorders) | 4 | 4 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 8 | 1 | 0
Nasopharyngitis (Infections and infestations) | 32 | 16 | 9
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 0
Gastritis (Gastrointestinal disorders) | 3 | 1 | 3
Hypertension (Vascular disorders) | 6 | 4 | 1
Nausea (Gastrointestinal disorders) | 6 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Gastroenteritis (Infections and infestations) | 7 | 0 | 1
Pharyngitis (Infections and infestations) | 6 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 18 | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.